CLINICAL TRIAL: NCT01985152
Title: A Placebo-Controlled, Phase I, Single-center Evaluation of the Single-dose Pharmacokinetics Study of Azilsartan Trimethylethanolamine
Brief Title: A Phase Ⅰa Study of Azilsartan Trimethylethanolamine in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: HS-AZTP1a
Record Dates: First submitted 2013-10-31; First posted 2013-11-15 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Health

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- 1.Azilsartan Trimethylethanolamine (Experimental): Single dose of Azilsartan Trimethylethanolamine with 8.75mg,orally
  Interventions: Drug: Azilsartan Trimethylethanolamine
- 2.Azilsartan Trimethylethanolamine (Experimental): Single dose of Azilsartan Trimethylethanolamine with 17.5mg,orally
  Interventions: Drug: Azilsartan Trimethylethanolamine
- 3.Azilsartan Trimethylethanolamine (Experimental): Single dose of Azilsartan Trimethylethanolamine with 35mg,orally
  Interventions: Drug: Azilsartan Trimethylethanolamine
- 4.Azilsartan Trimethylethanolamine (Experimental): Single dose of Azilsartan Trimethylethanolamine with 70mg,orally
  Interventions: Drug: Azilsartan Trimethylethanolamine
- 5.Azilsartan Trimethylethanolamine (Experimental): Single dose of Azilsartan Trimethylethanolamine with 140mg,orally
  Interventions: Drug: Azilsartan Trimethylethanolamine
- 6.Azilsartan Trimethylethanolamine (Experimental): Single dose of Azilsartan Trimethylethanolamine with 210mg,orally
  Interventions: Drug: Azilsartan Trimethylethanolamine
- 7.Azilsartan Trimethylethanolamine (Experimental): Single dose of Azilsartan Trimethylethanolamine with 280mg,orally
  Interventions: Drug: Azilsartan Trimethylethanolamine
- Placebo (Placebo Comparator): Placebo-matching tablets, orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azilsartan Trimethylethanolamine
  Arms: 1.Azilsartan Trimethylethanolamine; 2.Azilsartan Trimethylethanolamine; 3.Azilsartan Trimethylethanolamine; 4.Azilsartan Trimethylethanolamine; 5.Azilsartan Trimethylethanolamine; 6.Azilsartan Trimethylethanolamine; 7.Azilsartan Trimethylethanolamine
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the Pharmacokinetics and safety of Azilsartan Trimethylethanolamine in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females
* Aged from 18 years to 45 years
* Body mass index (BMI) 19 to 25kg/m2

Exclusion Criteria:

* Has a known sensitivity to angiotensin II receptor blocker（ARB）
* With evidence of uncontrolled renal, hepatic, central nervous system, respiratory, cardiovascular, or metabolic dysfunction, in the opinion of the investigator or medical monitor
* Has known or suspected history of alcoholism or drug abuse or misuse
* With a history of laboratory results that show the presence of hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCVAb), or human immunodeficiency virus (HIV)
* Pregnant,lactating，menstrual
* Vegetarian
* Postural hypotension
* Systolic blood pressure<100mmHg，or>130mmHg;and/or diastolic blood pressure<70mmHg,or>90mmHg

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2013-09; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
To study the Pharmacokinetics of Azilsartan Trimethylethanolamine by assessment of drug concentration through blood sample analysis | Pre-dose to 72 hours post-dosee
Number of participants with adverse reactions | Pre-dose to 72 hours post-dose
  The trial shoud be terminated ，if more than a third of participants had grade 2 or more than 2 adverse reactions based on Common Terminology Criteria for Adverse Events(CTCAE) Version 4.02

CONTACTS AND LOCATIONS:
Overall Officials: Jie Hou, Associate Chief Physician, Principal Investigator — TEDA International Cardiovascular Hospital
Locations (1):
- TEDA International Cardiovascular Hospital, Tianjin, China